CLINICAL TRIAL: NCT07311187
Title: The Quiet Quitting Phenomenon Among Healthcare Workers: an Observational Study
Brief Title: Quiet Quitting, Quality of Life, and Coping Strategies Among Healthcare Workers
Acronym: QQS
Status: Active, not recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Mattia Morri, PT, Istituto Ortopedico Rizzoli
Other Study IDs: 202/2025/Oss/IOR
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Well-being at Work
Keywords: Quiet Quitting; Health Personnel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health Workers: Nurses and allied health workers
  Interventions: Other: Quiet Quitting Scale

INTERVENTIONS:
Other: Quiet Quitting Scale — The Quiet Quitting scale (QQs) will be used to assess the phenomenon of silent resignation and to identify possible prognostic factors.

SUMMARY:
The purpose of the study is to investigate the psychological and physical well-being of healthcare professionals working at an orthopedic surgical hospital. In particular, we want to assess the presence and spread of a new work phenomenon called "quiet quitting," a phenomenon that has spread significantly in recent years in many work contexts.

DETAILED DESCRIPTION:
STUDY SETTING The study will be conducted within the hospital services of the Istituto Ortopedico Rizzoli (IOR). The central site in Bologna, the Rizzoli-Sicilia Department, and the Departments of Orthopaedics and Traumatology and Physical and Rehabilitation Medicine of the Rizzoli-Argenta site will be involved.

VARIABLES

To describe the sample of enrolled healthcare workers and to identify potential risk factors related to quiet quitting, the following variables will be collected in categorical form to ensure anonymity:

Age, classified into three categories: 18-30 years, 30-50 years, and >50 years

Sex

Educational level, classified into three categories: high school diploma, bachelor's degree, and postgraduate education

Profession (nurses, physiotherapists, technical area professionals, healthcare assistants)

Years of work experience (<5 years; 5-20 years; >20 years)

Years of employment at the enrolling hospital (<1 year; 1-5 years; >5 years)

Presence of minor children in the household (yes/no)

Presence of elderly parents in the family environment (yes/no)

Work activity involving night shifts (yes/no)

Work activity on public holidays (yes/no)

On-call duty (yes/no)

Holding a functional/managerial role (yes/no)

Area of work activity (inpatient wards; outpatient services; critical care units/services; technical services)

Correspondence between expectations and job assignment/work activity

In describing their work context, participants will also be asked to express their perceptions regarding the role of training, autonomy and staff recognition, career development opportunities, outcome monitoring, and communication. Each item will be rated on a 1-5 Likert scale, where 0 indicates a minimally relevant aspect and 5 a highly relevant aspect.

ENROLLMENT TIMELINE The estimated total duration of the study is 2 years from approval by the Ethics Committee. The enrollment period for the first data collection is planned from June 2025 to December 2025. The second data collection will be conducted during 2026.

SAMPLE SIZE AND STATISTICAL ANALYSIS A quality improvement project conducted at the Istituto Ortopedico Rizzoli on a sample of 76 nurses reported a quiet quitter prevalence of 46.6%. Assuming a 95% confidence level and a confidence interval width of 10%, the estimated sample size is at least 382 healthcare workers.

Collected data will be reported as mean and standard deviation or median and percentiles for continuous variables, according to their distribution, and as absolute and percentage frequencies for dichotomous/categorical variables. The group defined as "quiet quitters" will include workers reporting a score greater than 2.06 on the Quiet Quitting Scale. Variables will be described for the overall enrolled population and compared between quiet quitters and non-quiet quitters.

Identification of risk factors associated with the quiet quitter condition will be performed using univariate analyses, applying the chi-square test for dichotomous variables and Student's t-test or the Mann-Whitney test for continuous variables. Variables with a statistical significance level <0.157 in the univariate analysis will be included in the multivariable logistic regression model. Data from the first phase will be compared with those from the second year of data collection to assess trends in the overall phenomenon of disengagement.

ENROLLMENT PROCEDURE Informed consent and data collection will be carried out using the REDCap platform, which will be configured to ensure participant anonymity. The same procedure will be applied at both data collection time points (baseline administration and follow-up). On both occasions, feedback on the study results will be provided to all healthcare workers through staff meetings and the dissemination of summary tables and graphs. Participants may withdraw at any time before completing the questionnaires by simply not completing them.

DATA COLLECTION Study participants will be enrolled on a voluntary and anonymous basis. Data will be collected through an anonymous survey, completed electronically using the REDCap platform. A draft version of the questionnaire and the assessment scales to be used are attached to the documentation (see CRF). All workers will receive a dedicated participation link and will be able to complete the survey, which has an estimated duration of approximately 15 minutes, during working hours. Upon completion of data collection, data will be exported to an Excel file and stored in an electronic database for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* All workers in the healthcare sector, such as nurses, physical therapists, technical professionals, and social
* Healthcare workers employed by the services and departments of the facilities involved.
* Workers who express their willingness to participate in the study

Exclusion Criteria:

* Workers employed on temporary contracts or on contracts with third parties other than the hospital involved
* Workers who are absent from work for more than 3 months during the survey period, such as workers on maternity leave, long-term sick leave, or accident leave.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be conducted within the hospital services of the Istituto Ortopedico Rizzoli (IOR). The central site in Bologna, the Rizzoli-Sicilia Department, and the Departments of Orthopaedics and Traumatology and Physical and Rehabilitation Medicine of the Rizzoli-Argenta site will be involved.
Sampling Method: Non-Probability Sample
Enrollment: 382 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Quiet Quitting scale | The Quiet Quitting Scale survey was first conducted in June 2025 and will be repeated in 2026.
  The scale consists of nine items that investigate three main aspects of the phenomenon: detachment, understood as emotional separation from work-related concerns and thoughts; lack of motivation, understood as reduced drive to actively engage in one's work; and lack of initiative, understood as a low propensity to go beyond the minimum requirements of supervisors, i.e., to engage in non-mandatory activities. Responses to each item are provided on a 5-point Likert scale ranging from 1 to 5. The overall score on the scale is reported as the average of the items, and an average score above 2.06 identifies a 'quiet quitter', i.e. a person who experiences the phenomenon of silent abandonment.

SECONDARY OUTCOMES:
Quality of life (SF-12 scale) | The Quality of life survey was first conducted in June 2025 and will be repeated in 2026.
  The quality of life of healthcare workers will be measured using the Short-Form 12. The scale was designed to assess quality of life using 12 items with responses ranging from 2 to 6 levels. The overall score will be reported on two main dimensions: physical health and mental health. The score will be calculated in accordance with the manual proposed by the authors who validated the scale in Italian.
Mindfulness Organizing Scale (MOS) | The Mindfulness Organizing Scale survey was first conducted in June 2025 and will be repeated in 2026.
  The mindfulness and coping strategies implemented by professionals within the organization will be measured using the Mindfulness Organizing Scale (MOs). This scale consists of 9 items graded on a 3-point Likert scale (1 = not at all; 2 = somewhat; 3 = very much in agreement) with a score ranging from 9 to 27, with a higher score indicating better mindfulness strategies. The overall score will be reported as the average of the items completed.

CONTACTS AND LOCATIONS:
Overall Officials: Mattia Morri, Principal Investigator — IRCCS Istituto Ortopedico Rizzoli
Locations (1):
- SAITeR IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy, Italy

IPD SHARING:
Plan to Share IPD: No
data will be made available upon reasonable request to the Principal Investigator.

REFERENCES:
- [Result] Magnano, P., Platania, S., Ramaci, T., & Santisi, G. (2017). VALIDATION OF THE ITALIAN VERSION OF THE MINDFULNESS ORGANIZING SCALE (MOS) IN ORGANIZATIONAL CONTEXTS. 24(1).
- [Result] Apolone G, Mosconi P. The Italian SF-36 Health Survey: translation, validation and norming. J Clin Epidemiol. 1998 Nov;51(11):1025-36. doi: 10.1016/s0895-4356(98)00094-8. PMID 9817120
- [Result] Galanis, P., Katsiroumpa, A., Vraka, I., Konstantakopoulou, O., Moisoglou, I., Gallos, P., & Kaitelidou, D. (2023). Quiet quitting among employees: A proposed cut-off score for the "Quiet Quitting" Scale. Research Square. https://doi.org/10.21203/rs.3.rs-3076541/v1
- [Result] Galanis P, Katsiroumpa A, Vraka I, Siskou O, Konstantakopoulou O, Moisoglou I, Gallos P, Kaitelidou D. The quiet quitting scale: Development and initial validation. AIMS Public Health. 2023 Oct 17;10(4):828-848. doi: 10.3934/publichealth.2023055. eCollection 2023. PMID 38187899